CLINICAL TRIAL: NCT01508260
Title: Ultrafiltration (Aquapheresis) in the Management of Patients With Leukemia and Severe Fluid Overload
Brief Title: Ultrafiltration (Aquapheresis) in Patients With Leukemia and Severe Fluid Overload
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2011-0475
Record Dates: First submitted 2012-01-09; First posted 2012-01-11 (Estimated); Last update posted 2013-04-05 (Estimated); Status verified 2013-04

CONDITIONS: Leukemia
Keywords: Leukemia; Aquapheresis; Ultrafiltration; Aquadex pump; Severe Fluid Overload; Diuretic therapy; Dyspnea; Orthopnea; Paroxysmal nocturnal dyspnea; PND; Peripheral edema; Rales; Jugular venous distension; JVD; Hypoxia; Pulmonary edema by chest X-ray; Furosemide; Lasix
MeSH Terms: conditions — Leukemia; Edema; Dyspnea; Dyspnea, Paroxysmal; Respiratory Sounds; Hypoxia | interventions — Furosemide

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Pilot Phase Aquapheresis (Experimental): The first portion of this study is an open label pilot experience to evaluate the safety of aquapheresis in leukemia patients with severe fluid overload non-responsive to diuretics. A total of 10 patients will be treated.
  Interventions: Procedure: Aquapheresis
- Aquapheresis (Experimental): Participant connected to aquapheresis pump through an intravenous (IV) catheter placed in forearm. About 6 teaspoons of blood will flow through the blood circuit, and the excess fluid will slowly be collected in the collection bag. The exact length of time of aquapheresis treatment is determined by how much fluid needs to be removed and how fast it can be removed. The average treatment is about 24 hours but can extend up to 7 days. About 6 liters or 13 pounds will be removed.
  Interventions: Procedure: Aquapheresis
- Diuretics (Active Comparator): Furosemide by vein over about 15 minutes every 8 hours or by vein as a continuous (non-stop) infusion.
  Interventions: Drug: Furosemide

INTERVENTIONS:
Procedure: Aquapheresis — Participant connected to aquapheresis pump through an intravenous (IV) catheter placed in forearm. Average treatment is about 24 hours but can extend up to 7 days.
  Other Names: Aquadex pump
  Arms: Aquapheresis; Pilot Phase Aquapheresis
Drug: Furosemide — 20-40 mg by vein every 8 hours as indicated for optimal diuresis to achieve negative fluid balance or 0.5 to 5 mg per hour by continuous infusion.
  Other Names: Furomide; Lasix
  Arms: Diuretics

SUMMARY:
The goal of this clinical research study is to learn about the safety and level of effectiveness of aquapheresis compared to diuretic drugs. Diuretic drugs are designed to help the kidneys to form more urine. They also remove fluids from patients with severe fluid overload who have not responded to diuretics.

Aquapheresis is a procedure that removes excess fluid from the body. Blood containing too much salt and water is withdrawn from the body using catheters (sterile flexible tubes) and passed through a special filter. The filter separates the excess salt and water from the blood. The blood is returned to the patient and the fluid is collected in a bag to be disposed. Aquapherisis may benefit patients by removing excess fluid and salt from the body.

DETAILED DESCRIPTION:
Study Groups:

If you are found to be eligible to take part in this study, you will be assigned to a study group based on when you join this study. The first group of 10 participants to join the study will be enrolled in the Pilot portion of the study. The next group of up to 40 participants will be enrolled in the Randomized portion of the study.

In the Pilot portion of the study, researchers want to learn about the safety and level of effectiveness of aquapheresis in leukemia patients with severe fluid overload who do not respond to diuretics.

If you are in the Randomized portion of the study, you will be randomly assigned (as in the flip of a coin) to 1 of 2 groups. You will have an equal chance of being assigned to each group.

* Group A will receive aquapheresis.
* Group B will receive furosemide. The doctor will discuss this with you.

If you are in Group A, you will be connected to the aquapheresis pump through an intravenous (IV) catheter placed in your forearm. The pump looks like the ones used to infuse IV drugs. It will hang on a pole by your bed. About 6 teaspoons of your blood will flow through the blood circuit, and the excess fluid will slowly be collected in the collection bag. The exact length of time of aquapheresis treatment is determined by how much fluid needs to be removed and how fast it can be removed. The average treatment is about 24 hours but can extend up to 7 days. About 6 liters or 13 pounds will be removed.

If you are in Group B, you will receive one of the following for as the doctor thinks it is needed (until most of the excess fluid is removed):

* furosemide by vein over about 15 minutes every 8 hours
* furosemide by vein as a continuous (non-stop) infusion

Both Groups:

If the doctor thinks it is needed, you will be given other standard of care drugs such as albumin and metolazone to help your kidneys to make more urine. The study staff will tell you about these drugs, how they will be given, and the possible risks.

Study Visits:

Every day while you are receiving aquapheresis or diuretic treatment:

* You will be asked about any symptoms you may be having.
* You will have a physical exam, including measurement of your vital signs (blood pressure, heart rate, and breathing rate) and weight.
* You will be asked how much you drank. The study staff will measure how much you urinate.
* Your leg will be measured for swelling due to fluid retention.

At least every other day, blood (about 4 teaspoons) will be drawn for routine tests.

If the doctor thinks it is needed, you will have a chest x-ray on Day 3.

Length of Participation:

If you are in Group A, you will remain on study treatment for as long as the doctor thinks it is needed (possibly about 1-7 days).

If you are in Group B, you will receive standard treatment for as long as your doctor thinks it is needed.

You will no longer be able to receive the study treatment (Group A) or you will be taken off study (Group B) if intolerable side effects occur or if you are unable to follow study directions.

Your participation on the study will be over once you have completed the end-of-study follow-up visit.

End-of-Treatment Visit:

After you stop taking the study treatment or standard treatment, the following tests and procedures will be performed:

* You will be asked about any symptoms you may be having.
* You will have a physical exam, including measurement of your vital signs and weight.
* You will be asked how much you drank. The study staff will measure how much you urinate.
* Your leg will be measured for swelling due to fluid retention.
* Blood (about 4 teaspoons) will be drawn for routine tests.
* If the doctor thinks it is needed, you will have a chest x-ray.

End-of-Study Follow-up Visit:

At 30 days after the end of study therapy:

* You will have a physical exam, including measurement of your vital signs and weight.
* You will be asked about any symptoms you may be having.
* Your leg will be measured for swelling due to fluid retention.

This is an investigational study. The Aquadex FlexFlow™ Fluid Removal Systems pump used for aquapheresis is FDA approved and commercially available for patients with fluid overload. Using the Aquadex FlexFlow™ Fluid Removal Systems pump in patients with leukemia to remove excess fluid is investigational. Furosemide is FDA approved and commercially available for other uses such as the treatment of swelling caused by heart failure or kidney or liver problems.

Up to 50 patients will be enrolled in this study. All will be enrolled at MD Anderson.

ELIGIBILITY:
Inclusion Criteria:

1. All patients must be 18 years of age or older and have a diagnosis of leukemia and be hospitalized on leukemia floor or MICU
2. Weight gain of 10 pounds or more.
3. In addition, patients should have 2 or more signs and symptoms of fluid overload such as: dyspnea, orthopnea, paroxysmal nocturnal dyspnea (PND), peripheral edema, rales, jugular venous distension (JVD), hypoxia (pulse ox < 90% on room air) and pulmonary edema by chest X-ray.
4. AND be poorly responsive to diuretics defined as positive fluid balance or < 1% decrease in current body weight / 24 hours with use of furosemide 60 mg IV/24h.
5. Subjects will be eligible regardless of poor performance, organ dysfunctions, organ failures, or other criteria of decompensation and/or debilitation.
6. Subjects will be eligible regardless of platelet counts.
7. Patients may be on a regular floor or in the intensive care unit.
8. They may be on respiratory mechanical ventilation or not.

Exclusion Criteria:

1. Indication for dialysis (as judged necessary by nephrology (hyperkalemia, acidosis).
2. AKI defined as 100% increase in baseline creatinine.
3. Hypotension (SBP < 90mmHg).
4. Pregnant or breastfeeding women are excluded.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2013-03; Primary Completion 2018-03 (Estimated)

PRIMARY OUTCOMES:
Safety and Efficacy of Aquapheresis versus Diuretic Therapy | 72 hours
  Primary end point is success rate defined as achievement of weight loss of 7 pounds or 50% of weight gain, whichever is greater without >/=100% increase of baseline creatinine at 72 hours.

SECONDARY OUTCOMES:
Complete Response | 72 hours
  Complete response defined as achievement of 80% removal of fluid overload compared to dry body weight (average body weight before being sick and hospitalized) without ≥100% increase of baseline creatinine at 72 hours.

CONTACTS AND LOCATIONS:
Overall Officials: Gloria Iliescu, MD, Principal Investigator — UT MD Anderson Cancer Center

REFERENCES:
- See also: UT MD Anderson Cancer Center Website — http://www.mdanderson.org